CLINICAL TRIAL: NCT02632331
Title: Pharmacokinetic (PK) Study of ASP8825 - Evaluation of the Effect of Food on the Pharmacokinetics
Brief Title: ASP8825 - A Study to Investigate the Food Effect on the Pharmacokinetics of ASP8825
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 8825-CL-0014
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Volunteers
Keywords: Food effect; Pharmacokinetics; ASP8825; XP13512
MeSH Terms: interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasted dosing preceding group (Experimental)
  Interventions: Drug: ASP8825
- Fed dosing preceding group (Experimental)
  Interventions: Drug: ASP8825

INTERVENTIONS:
Drug: ASP8825 — Oral
  Other Names: gabapentin enacarbil

SUMMARY:
The objective of this study is to evaluate the effect of food on the pharmacokinetics and safety after administration of ASP8825 in healthy non-elderly adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: ≥50.0 kg and <80.0 kg
* Body mass index BMI: ≥17.6 and <26.4 [BMI= Body weight (kg)/(Height (m))2]

Exclusion Criteria:

* Subjects who received any study drugs in other clinical trials or post-marketing studies within 120 days before screening
* Subjects who received or are scheduled to receive medications (including over-the-counter [OTC] drugs) within seven days before the hospital admission day of period 1.
* Subjects who deviate from the normal range of blood pressure, pulse rate, body temperature and standard 12-lead ECG at screening or the hospital admission day of period 1
* Subjects who meet any of the criteria for laboratory tests at screening or the hospital admission day of period 1. Normal ranges of each test specified at the study site or the test/assay organization will be used as the normal ranges in this study.
* Subjects with a complication of drug allergies
* Subjects who developed upper gastrointestinal symptoms (e.g., nausea, vomiting, and stomachache) within seven days before the hospital admission day of period 1
* Subjects with a complication or history of hepatic disease (hepatitis viral and drug-induced liver injury, etc.)
* Subjects with a complication or history of heart disease (cardiac failure congestive, angina pectoris and arrhythmia requiring treatments, etc.)
* Subjects with a complication or history of respiratory disease (severe asthma bronchial and bronchitis chronic, etc.) (except for a history of non-severe infantile asthma)
* Subjects with a complication or history of alimentary disease (severe peptic ulcer, reflux esophagitis, etc.) (except for a history of appendicitis)
* Subjects with a complication or history of renal disease (acute kidney injury, glomerulonephritis, nephritis interstitial, etc.) (except for a history of calculus)
* Subjects with a complication or history of cerebrovascular disorder (cerebral infarction, etc.)
* Subjects with a complication or history of malignant tumor
* Subjects who have a habit of excessive alcohol drinking or smoking
* Subjects who previously received administration of ASP8825

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameter of gabapentin: Cmax | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36 and 48 hr after dosing
  Cmax: Maximum concentration
PK parameters of gabapentin: AUClast | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36 and 48 hr after dosing
  AUClast: Area under the concentration-time curve from the time of dosing extrapolated to the last measurable concentration
Safety assessed by AEs | Up to 8 days after the final study drug dosing
  AEs: Adverse Events
Safety assessed by Vital signs | Up to 3 days after the each study drug dosing
  Supine blood pressure, supine pulse rate and axillary body temperature
Safety assessed by Laboratory tests | Up to 3 days after the each study drug dosing
  Hematology, blood biochemistry, and urinalysis
Safety assessed by 12-lead ECGs | Up to 3 days after the each study drug dosing
  ECG: Electrocardiogram

SECONDARY OUTCOMES:
PK parameters of gabapentin tmax | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36 and 48 hr after dosing
  tmax: Time of Cmax
PK parameter of gabapentin: AUCinf | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36 and 48 hr after dosing
  AUCinf: Area under the concentration-time curve from the time of dosing extrapolated to time infinity
PK parameters of gabapentin: t1/2 | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36 and 48 hr after dosing
  t1/2: Terminal elimination half-life
PK parameters of gabapentin: CL/F | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36 and 48 hr after dosing
  CL/F: Apparent total systemic clearance
PK parameters of gabapentin: MRTinf | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36 and 48 hr after dosing
  MRTinf: Mean residence time from the time of dosing extrapolated to time infinity
PK parameters of gabapentin: MRTlast | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36 and 48 hr after dosing
  MRTlast: Mean residence time from the time of dosing extrapolated to the last measurable concentration
PK parameters of gabapentin: kel | Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36 and 48 hr after dosing
  kel: Terminal elimination rate constant

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Undecided